CLINICAL TRIAL: NCT03476746
Title: Dermatopharmacokinetic Trial of LEO 90100 Foam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LP0053-1417
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2018-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A single application of LEO 90100 foam and Dovobet® ointment will be applied to multiple test sites on the innerside of both arms of trial subjects. The trial consists of 2 parts. The first part, (pilot part) will evaluate the pharmacokinetic profile of LEO 90100 foam and Dovobet® ointment by measuring the amount of each of the active ingredients in the stratum corneum and determine conditions for the second part of the trial. The second part (pivotal part) will compare the amount of each of the active ingredients at steady state or close-to-steady state between LEO 90100 foam and Dovobet® ointment. The sample size and the number of application sites in the pivotal part will be determined based on the results of the pilot part.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEO 90100 foam (Experimental): LEO 90100 foam (containing calcipotriol hydrate 52.2 µg/g [equivalent to 50.0 µg/g calcipotriol] plus betamethasone dipropionate 0.643 mg/g).
  Pilot part: 6 single applications of LEO 90100 foam on Day 1 (for 12 sites in total).
  Pivotal part: To be decided based on the result of the pilot part
  Interventions: Drug: LEO 90100 foam
- Dovobet® ointment (Active Comparator): Pilot part: 6 single applications of Dovobet® ointment on Day 1 (for 12 sites in total).
  Pivotal part: To be decided based on the result of the pilot part
  Interventions: Drug: Dovobet® ointment

INTERVENTIONS:
Drug: LEO 90100 foam — A foam formulation of the active comparator Dovobet® ointment
  Arms: LEO 90100 foam
Drug: Dovobet® ointment — Ointment formulation containing same active ingredients as LEO 90100 foam
  Arms: Dovobet® ointment

SUMMARY:
This is a phase 1, single centre trial in Japanese healthy male subjects comparing the amount of active ingredients of LEO 90100 foam and Dovobet® ointment in the stratum corneum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male subjects, aged 20 to 40 years inclusive

Exclusion Criteria:

* Body Mass Index outside the range 18-25 kg/m²
* Use of any medication (systemic or topical) within 2 weeks of Day 1.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
The amount of each of the 2 active ingredients, calcipotriol and betamethasone dipropionate, in the stratum corneum obtained by means of tape stripping after application of LEO 90100 foam and Dovobet® ointment. | 2, 4, 6, 8, 12 and 24 hr after drug application.
  Amount (nanogram) of calcipotriol and betamethasone dipropionate in the stratum corneum will be compared between the two formulations by selected time points using an ANOVA model with treatment/formulation as systematic effect.

SECONDARY OUTCOMES:
Safety data - number of adverse events | up to 15 Days after drug application
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (1):
- Investigational site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No